CLINICAL TRIAL: NCT03425422
Title: Autonomic Regulation Therapy to Enhance Myocardial Function and Reduce Progression of Heart Failure With Reduced Ejection Fraction
Brief Title: ANTHEM-HFrEF Pivotal Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company decision to stop enrolling not associated with any safety concerns.
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-07
Record Dates: First submitted 2018-01-26; First posted 2018-02-07 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure; Heart Failure, Congestive; Heart Failure, Systolic
Keywords: Vagus nerve stimulation
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Therapy (Experimental): VITARIA system implantation on the right cervical vagus nerve in addition to stable guideline-directed medical therapy
  Interventions: Device: VITARIA System
- Control (No Intervention): Stable guideline-directed medical therapy

INTERVENTIONS:
Device: VITARIA System — Chronic stimulation of the right cervical vagus nerve
  Arms: Therapy

SUMMARY:
A multi-center randomized controlled clinical trial to evaluate Autonomic Regulation Therapy with the VITARIA system in patients with symptomatic heart failure and reduced ejection fraction.

DETAILED DESCRIPTION:
ANTHEM-HFrEF is a multi-center, open-label, randomized controlled clinical trial with an adaptive design. Patients with symptomatic heart failure and reduced LVEF will be enrolled and randomized 2:1 to receive VITARIA system implantation on the right cervical vagus nerve in addition to stable guideline-directed medical therapy (therapy), or to continue receiving stable guideline-directed medical therapy alone (control arm).

Subjects in the therapy arm will receive continuous, periodic VNS stimulation after surgery is completed, and will undergo visits for VNS up titration over a period of 3 months. Subjects in the control arm will also undergo scheduled visits at a similar frequency as the titration visits that are scheduled for subjects in the therapy arm. Data for safety and efficacy assessments will be collected for both study arms at 4 weeks post-randomization, every 3 months for the first 12 months, and every 4 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above
2. Willing and capable of providing informed consent
3. Capable of participating in all testing associated with this clinical investigation
4. Stable, guideline-directed medical therapy for at least 4 weeks before subject screening. Unrestricted changes in diuretics are allowed during the 4 weeks, as long as the subject remains on a diuretic. If the use of an ARNI is being contemplated for a study subject, ARNI should be administered, and GDMT optimized, before the subject is randomized. No more than a 100% increase or 50% decrease of the dosage of any medication other than a diuretic is permitted. For these medications, medication changes within a class are allowed, as long as the equivalent dosage is within these specified limits
5. Stable symptomatic heart failure NYHA class III; or NYHA class II with a heart failure hospitalization in the previous 12 months. HF hospitalization may include an overnight hospital or hospital-based observation unit stay with a primary diagnosis of HF, or an emergency department visit with a primary diagnosis of HF, and will in either case include documentation of intravenous HF therapy administration or other intervention for HF
6. Left ventricular ejection fraction (EF) ≤ 35% and left ventricular end-diastolic diameter (LVEDD) < 8.0 cm, as confirmed by the core echocardiography laboratory during screening
7. N-terminal pro-BNP (NT-proBNP) level of at least 800 pg/mL, as determined by the core laboratory; or NT-proBNP level of at least 1200 pg/mL, as determined by the core laboratory, for patients with permanent atrial fibrillation or reporting signs or symptoms of atrial fibrillation at the time that the NT-proBNP sample is drawn
8. Received a standard cardiac assessment, including history, physical exam, and electrocardiogram, and determined by a heart failure cardiologist and study surgeon to be an appropriate candidate for the study's surgical procedure
9. Physically capable and willing to perform repeated 6-minute walk tests associated with the study, and having a baseline distance of between 150 and 450 meters. Symptoms limiting the duration of the 6 minute walk test must be due primarily to heart failure

Exclusion Criteria:

1. Refractory symptomatic hypotension (systolic blood pressure below 80 mmHg)
2. Complete AV block treated with unipolar pacemaker therapy
3. Currently implanted vagus nerve stimulation (VNS) device, baroreceptor activation therapy (BAT) device, other nerve stimulator, artificial or donor heart, or ventricular assist device (VAD)
4. Heart failure of non-ischemic origin for less than 6 months, or due to congenital heart disease, hypertrophic obstructive cardiomyopathy, or infiltrative cardiomyopathy (e.g. amyloidosis, sarcoidosis)
5. Moderate (3+) or severe (4+) aortic valve or mitral valve stenosis; moderate (3+) or severe (4+) aortic valve insufficiency; or severe (4+) mitral valve insufficiency
6. Symptomatic uncontrolled bradycardia
7. On renal dialysis
8. Involvement in any concurrent clinical study with an investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Event-free rate | 90 days
  The event-free rate, through 90 days after VITARIA implantation, from all VITARIA system-related and VITARIA implantation-related serious adverse events, as adjudicated by the Clinical Events Committee
Cardiovascular mortality and HF hospitalization | Through study completion, an average of 2 years
  A composite of cardiovascular mortality or heart failure hospitalization, as adjudicated by the Clinical Events Committee, based on time to first event after randomization

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - University of Alabama, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - Long Beach Memorial Hospital, Long Beach, California
  - Greater Los Angeles VA Medical Center, Los Angeles, California
  - Hartford Hospital, Hartford, Connecticut
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - UnityPoint Health - Methodist Hospital, Peoria, Illinois
  - Indiana University Health Ball Memorial Hospital, Muncie, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Medical Center, Burlington, Massachusetts
  - Michigan Heart, PC, Ypsilanti, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mount Sinai School St. Luke's, New York, New York
  - MetroHealth System, Cleveland, Ohio
  - ProMedica Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Penn State Health Milton Hershey Medical Center, Hershey, Pennsylvania
  - Pinnacle Health, Wormleysburg, Pennsylvania
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Premchand RK, Sharma K, Mittal S, Monteiro R, Dixit S, Libbus I, DiCarlo LA, Ardell JL, Rector TS, Amurthur B, KenKnight BH, Anand IS. Autonomic regulation therapy via left or right cervical vagus nerve stimulation in patients with chronic heart failure: results of the ANTHEM-HF trial. J Card Fail. 2014 Nov;20(11):808-16. doi: 10.1016/j.cardfail.2014.08.009. Epub 2014 Sep 1. PMID 25187002
- [Background] Premchand RK, Sharma K, Mittal S, Monteiro R, Dixit S, Libbus I, DiCarlo LA, Ardell JL, Rector TS, Amurthur B, KenKnight BH, Anand IS. Extended Follow-Up of Patients With Heart Failure Receiving Autonomic Regulation Therapy in the ANTHEM-HF Study. J Card Fail. 2016 Aug;22(8):639-42. doi: 10.1016/j.cardfail.2015.11.002. Epub 2015 Nov 11. PMID 26576716
- [Derived] Konstam MA, Udelson JE, Butler J, Klein HU, Parker JD, Teerlink JR, Wedge PM, Saville BR, Ardell JL, Libbus I, DiCarlo LA. Impact of Autonomic Regulation Therapy in Patients with Heart Failure: ANTHEM-HFrEF Pivotal Study Design. Circ Heart Fail. 2019 Nov;12(11):e005879. doi: 10.1161/CIRCHEARTFAILURE.119.005879. Epub 2019 Nov 14. PMID 31722536
- See also: ANTHEM-HFrEF Study Site — http://www.artforheartfailure.com